CLINICAL TRIAL: NCT03710512
Title: Evaluation of Early Relapse After Mandibular Lengthening Surgery With or Without the Use of a Bone Graft Substitute at the Osteotomy Site.
Brief Title: Evaluation of Early Relapse After Mandibular Lengthening Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Universitair Ziekenhuis Brussel (Other)
Responsible Party: Principal Investigator, Veerle Van Mossevelde, Datanurse, Universitair Ziekenhuis Brussel
Other Study IDs: EARLY RELAPSE AFTER MANDIBULAR
Record Dates: First submitted 2018-06-28; First posted 2018-10-18 (Actual); Last update posted 2018-10-18 (Actual); Status verified 2018-10

CONDITIONS: Mandibular Hypoplasia; Relapse
Keywords: hydroset
MeSH Terms: conditions — Micrognathism; Recurrence

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hydroset: patients receiving hydroset at osteotomy site
  Interventions: Procedure: Bilateral sagittal split osteotomy
- Control: patients not receiving hydroset at osteotomy site
  Interventions: Procedure: Bilateral sagittal split osteotomy

INTERVENTIONS:
Procedure: Bilateral sagittal split osteotomy — Bilateral sagittal split osteotomy of the mandible is a surgical procedure used to correct dentofacial discrepancies

SUMMARY:
The goal of this study is to evaluate whether the use of a bone graft substitute at the osteotomy site will result in better stability and diminish early relapse after mandibular lengthening surgery.

The study focuses on the evaluation of the following hypothesis:

The use of bone graft substitute at the osteotomy site has an influence on:

* The 3-dimensional stability of the osteotomy site
* Early relapse based in the plasticity of the site

DETAILED DESCRIPTION:
Bilateral sagittal split osteotomy (BSSO)of the mandible is a surgical procedure used to correct dentofacial discrepancies. Post-operative stability is of great concern for CMF (Cranio maxillo facial) surgeons as the goal is to achieve optimal functional outcomes, good aesthetic results and satisfaction of patients' concerns. Skeletal relapse is a known complication of mandibular lengthening surgery and is divided into two groups; short term or early relapse and long term or late relapse.

Short term relapse occurs within the first 6 to 8 weeks post-operatively and is due to intersegmental movement at the osteotomy site (osteotomy slippage) and osteosynthesis slippage. Late relapse is thought to be caused by progressive condylar resorption, a clinical entity affecting the temporomandibular joint.

The rationale to reconstruct the lateral cortical defect resulting from mandibular advancement with BSSO with a bone graft substitute lies in the prevention of an unaesthetic notching at the inferior border. The use of a self-hardening, space-occupying paste could add mechanical stability, thus increase 3D-stability at the osteotomy site and prevent early relapse.

The use of cone-beam computed tomography (CBCT) in the treatment planning and postoperative follow-up of orthognathic patients has provided the surgeons with a new three-dimensional imaging modality to evaluate the postoperative skeletal relapse and postoperative morphologic changes of the condyles. Skeletal relapse, as well as positional and dimensional changes of the condyles, can be quantified in three dimensions.

ELIGIBILITY:
Inclusion Criteria:

* Class II occlusion of non-syndromic origin, mandibular hypoplasia
* Availability of pre- and postoperative CBCT scans of sufficient quality
* Age: >10years

Exclusion Criteria:

* Previous orthognathic surgical treatment
* Simultaneously performed genioplasty
* Plate osteosynthesis
* Buccal plate fracture during surgery

Ages: 10 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Class II occlusion of non-syndromic origin, mandibular hypoplasia
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2018-09-11 (Actual); Primary Completion 2019-09-01 (Estimated); Study Completion 2019-12-30 (Estimated)

PRIMARY OUTCOMES:
early relapse by means of three dimensional color maps (CBCT) | the first 6 months postoperatively
  evaluation at the osteotomy gap, the position of the condyles, rami and chin

SECONDARY OUTCOMES:
condylar resorption by means of three dimensional color maps (CBCT) | the first 6 months postoperatively
  a three-dimensional volumetric analysis of the condylar head and the glenoid cavity

CONTACTS AND LOCATIONS:
Overall Officials: Erica Coppey, MD, Principal Investigator — Universitair Ziekenhuis Brussel; Maurice Mommaerts, Prof. Mult, Study Director — Universitair Ziekenhuis Brussel
Locations (1):
- Universitair Ziekenhuis Brussel, Jette, Vlaams Brabant, Belgium